CLINICAL TRIAL: NCT04295343
Title: Three-dimensional Rectal Water Contrast Transvaginal Ultrasonography Versus Computed Colonography in the Diagnosis of Rectosigmoid Endometriosis
Brief Title: Three-dimensional (3D) Rectal Water Contrast Transvaginal Ultrasonography Versus Computed Colonography in the Diagnosis of Rectosigmoid Endometriosis
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: 3dETV-CTC-ENDO
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Endometriosis, Sigmoid; Endometriosis, Rectum
Keywords: Rectosigmoid endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Colonography, Computed Tomographic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspicious of rectosigmoid endometriosis
  Interventions: Diagnostic Test: Three-dimensional (3D) rectal water contrast transvaginal ultrasonography; Diagnostic Test: Computed colonography

INTERVENTIONS:
Diagnostic Test: Three-dimensional (3D) rectal water contrast transvaginal ultrasonography — Rectal water contrast transvaginal ultrasonography is based on the distention of rectosigmoid with saline solution. Three-dimensional reconstructions convert standard 2D grayscale ultrasound acquisitions into a volumetric dataset.
Diagnostic Test: Computed colonography — Computed colonography or virtual colonoscopy uses special x-ray equipment to examine the large intestine. During the exam, a small tube is inserted a short distance into the rectum to allow for inflation with gas while computed tomographic images of the colon and the rectum are taken.

SUMMARY:
Rectosigmoid involvement by endometriosis causes intestinal symptoms such as constipation, diarrhea, and dyschezia. A non-invasive diagnosis of bowel endometriosis is relevant to provide the patients information on the potential hormonal or surgical treatments. The objective of the current study was to compare the performance of three-dimensional rectal water contrast transvaginal ultrasonography (3D-RWC-TVS) and computed colonography (CTC) in predicting the presence and characteristics of rectosigmoid endometriosis.

ELIGIBILITY:
Inclusion Criteria:

- pain and intestinal symptoms suggestive of rectosigmoid endometriosis

Exclusion Criteria:

* previous surgical diagnosis of intestinal endometriosis
* previous radiological diagnosis of intestinal endometriosis (based on Magnetic Resonance or double-contrast barium enema
* history of colorectal surgery (except appendectomy)
* contraindications to bowel preparation or computed colonography (such as non-- compliant patients and rectal malformations)
* previous bilateral ovariectomy
* psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinical presentation suspected for rectosigmoid endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
To compare the accuracy of 3D-RWC-TVS and CTC in the diagnosis of rectosigmoid endometriosis. | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.

SECONDARY OUTCOMES:
To compare the precision of 3D-RWC-TVS and CTC in estimating the length (mid-sagittal diameter) of the rectosigmoid endometriotic nodules | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.
To compare the accuracy of 3D-RWC-TVS and CTC in the diagnosis of multifocal rectosigmoid endometriosis. | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.
To compare the precision of 3D-RWC-TVS and CTC in estimating and the distance between the lower margin of the rectosigmoid endometriotic nodules and the anal verge | At maximum 6 months before laparoscopic surgical approach
  The results of imaging will be compared with surgical and histological findings.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, MD, PhD, Study Director — IRCCS Ospedale Policlinico San Martino
Locations (1):
- Ospedale Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrero S, Biscaldi E, Vellone VG, Venturini PL, Leone Roberti Maggiore U. Computed tomographic colonography vs rectal water- contrast transvaginal sonography in diagnosis of rectosigmoid endometriosis: a pilot study. Ultrasound Obstet Gynecol. 2017 Apr;49(4):515-523. doi: 10.1002/uog.15905. PMID 26935873
- [Background] Morotti M, Ferrero S, Bogliolo S, Venturini PL, Remorgida V, Valenzano Menada M. Transvaginal ultrasonography with water-contrast in the rectum in the diagnosis of bowel endometriosis. Minerva Ginecol. 2010 Jun;62(3):179-85. English, Italian. PMID 20595942
- [Result] Barra F, Biscaldi E, Scala C, Lagana AS, Vellone VG, Stabilini C, Ghezzi F, Ferrero S. A Prospective Study Comparing Three-Dimensional Rectal Water Contrast Transvaginal Ultrasonography and Computed Tomographic Colonography in the Diagnosis of Rectosigmoid Endometriosis. Diagnostics (Basel). 2020 Apr 24;10(4):252. doi: 10.3390/diagnostics10040252. PMID 32344709